CLINICAL TRIAL: NCT03835442
Title: A Placebo Controlled Trial With Baclofen for the Treatment of GERD Patients With Incomplete PPI Response
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Prof Dr Jan Tack, professor, Universitaire Ziekenhuizen KU Leuven
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: S51996
Record Dates: First submitted 2019-02-04; First posted 2019-02-08 (Actual); Last update posted 2019-02-08 (Actual); Status verified 2019-02

CONDITIONS: Gastro Esophageal Reflux
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Baclofen

STUDY DESIGN:
Intervention Model Description: randomized, parallel, double-blind, placebo-controlled, out-patient, single-center study
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- baclofen arm (Active Comparator): baclofen 10mg tid for 4 weeks
  Interventions: Drug: Baclofen
- placebos arm (Placebo Comparator): placebo tid for 4 weeks
  Interventions: Other: Placebos

INTERVENTIONS:
Drug: Baclofen — baclofen 10mg tid for 4 weeks
  Other Names: Lioresal
  Arms: baclofen arm
Other: Placebos — placebo tid for 4 weeks
  Arms: placebos arm

SUMMARY:
Reflux (acid and non-acid) mainly occurs during transient LES relaxations (TLESRs). The gamma-aminobutyric acid (GABA) receptor type B agonist baclofen was shown to inhibit TLESRs, thereby significantly decreasing acid reflux after a meal in healthy controls and in patients with GERD.

The primary objective of this study is to assess the efficacy (assessed by reflux symptom questionnaire and pH-impedance recordings) of baclofen 10mg three times daily vs. placebo in GERD patients with an incomplete response to PPI therapy.

The secondary objective is to assess the predictive value of reflux assessment (by pH-impedance recordings) on the primary outcome.

DETAILED DESCRIPTION:
This is a randomized, parallel, double-blind, placebo-controlled, out-patient, single-center study. Eligible subjects will be randomly assigned to receive either oral baclofen 10 mg or placebo t.i.d for a period 4 weeks. After 4 weeks all patients will be given the standard dose of baclofen 10 mg t.i.d. (open label), for another 4 weeks. The b.i.d. PPI therapy will be continued for the entire study duration.

Approximately 90 evaluable subjects with typical GERD symptoms (heartburn and/or regurgitation) will participate in this study and will be randomized on a 1:1 basis: 45 subjects each will be in the placebo and baclofen 10 mg three times daily group. Subjects will be considered to have completed the study if they complete the week 4 visit.

Medication will consist of identically-looking capsules of baclofen or placebo. Patients will take 1 capsule containing 5 mg baclofen with meals t.i.d for 7 days and then 1 capsule containing 10 mg baclofen with meals t.i.d for the remaining 21 days.

Prior to visit 1, all subjects included in the study will undergo a 24 hr pH-impedance study which was requested by the treating physician. This investigation is part of the standard clinical work up and will not be part of the study protocol.

Informed consent is to be signed and dated by the subject before any study related procedures are performed. The date of each visit to the clinic and the date and time of the last dose of test article will be recorded.

Throughout the study patients will be asked to complete daily a short questionnaire (ReQuest) for reflux symptoms.

ELIGIBILITY:
Inclusion Criteria:

* 18 - 75 years old
* History of typical (heartburn/regurgitation) or atypical GERD symptoms during PPI treatment, at least 3 times per week for 12 weeks. Daily intake of PPI treatment 12 weeks prior to inclusion.
* Sexually active women of child bearing potential participating in the study must use a medically acceptable form of contraception. Medically acceptable forms of contraception include oral contraceptives, injectable or implantable methods, intrauterine devices, or properly used barrier contraception.
* Subjects must be capable of understanding and be willing to provide signed and dated written voluntary informed consent before any protocol-specific screening procedures are performed.

Exclusion Criteria:

* Endoscopic signs of severe erosive esophagitis (≥ grade C, Los Angeles classification) on endoscopy performed during PPI treatment in the 6 months prior to screening.
* Systemic diseases, known to affect esophageal motility.
* Surgery in thorax or in the upper part of the abdomen.
* Treatment with baclofen prior to the start of the study.
* Regular use of medications such as: anticholinergics, tricycle antidepressants.
* Significant neurological, respiratory, hepatic, renal, haematological, cardiovascular, metabolic or gastroinestinal cerebrovascular disease as judged by the investigator
* Absence of PPI intake for at least 2 consecutive days in the 2 weeks prior to the screening.
* Pregnancy or breast feeding.
* History of poor compliance. History of/or current psychiatric illness that would interfere with ability to comply with protocol requirements or give informed consent. (well-compensated depression is allowed).
* History of alcohol or drug abuse that would interfere with ability to comply with protocol requirements.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-01 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
efficacy of baclofen on reflux symptom questionnaire | Change from baseline in ReQuest scores at 4 weeks
  To assess the effect of baclofen on reflux symptom questionnaire by ReQuest
efficacy of baclofen on pH-impedance recordings | Change from baseline in reflux parameters (total number of reflux episodes) on 24h pH-impedance monitoring at 4 weeks
  To assess of baclofen on 24 hour pH-impedance recordings

SECONDARY OUTCOMES:
Predictive value of the reflux monitoring | Is SAP at baseline predictor of response at 4 weeks
  To assess the predictive value of the 24 hour pH-impedance monitoring (symptom association probability = SAP) on the primary outcome

CONTACTS AND LOCATIONS:
Overall Officials: Jan Tack, PhD, MD, Principal Investigator — UZ Leuven

IPD SHARING:
Plan to Share IPD: No